CLINICAL TRIAL: NCT05305274
Title: The Effect of Age and Refraction in Predicting Myopia Progression With Risk Under COVID-19 in a 3-year Follow-up of a Chinese Cohort
Brief Title: Age and Refraction in Predicting Myopia Progression in COVID-19
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022018
Record Dates: First submitted 2022-03-29; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Refraction Error; Myopia
MeSH Terms: conditions — Refractive Errors; Myopia | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 2019 screening: 34,400 schoolchildren with a 36-month follow-up from 2019 to 2021.
  Interventions: Other: screening
- 2020 screening: 34,400 schoolchildren with a 36-month follow-up from 2019 to 2021.
  Interventions: Other: screening
- 2021 screening: 34,400 schoolchildren with a 36-month follow-up from 2019 to 2021.
  Interventions: Other: screening

INTERVENTIONS:
Other: screening — This study included 34,400 students, as part of the Tianjin Eye Study who performed a 3-year follow-up from 2019 to 2021. All participants underwent yearly noncycloplegic refraction and ocular examinations. Time-related changes in sphere, cylinder, and spherical equivalent (SE) measurements in both sexes were analyzed.

SUMMARY:
To determine the longitudinal changes of age and refraction in predicting myopia progression with risk under the coronavirus disease 2019 (COVID-19) pandemic in a 3-year follow-up of a Chinese cohort.

DETAILED DESCRIPTION:
This was part of the large-scale Tianjin Eye Study, a population-based cohort study that longitudinally investigates the relationship between the age, refraction, and development of childhood RE in Tianjin, China.

ELIGIBILITY:
Inclusion Criteria:

* no concurrent eye disease;
* age 6-15 years.

Exclusion Criteria:

* significant systemic illnesses
* ocular conditions that could affect the corneal curvature, including congenital corneal diseases,
* pterygium, keratoconus, other corneal degeneration or dystrophy conditions,
* media opacity, uveitis, glaucoma
* a history of intraocular surgery, refractive surgery,
* neurologic or retinal diseases, current corneal refractive therapy (ortho-K),
* low-dose atropine therapy for myopia control

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study includes 34,400 schoolchildren, with a 36-month follow-up from 2019 to 2021. In addition to RE considerations, the inclusion criteria were: no concurrent eye disease; age 6-15 years. The exclusion criteria were: significant systemic illnesses or ocular conditions that could affect the corneal curvature, including congenital corneal diseases, pterygium, keratoconus, other corneal degeneration or dystrophy conditions, media opacity, uveitis, glaucoma or a history of intraocular surgery, refractive surgery, neurologic or retinal diseases, current corneal refractive therapy (ortho-K), or low-dose atropine therapy for myopia control. The ethics board of the Tianjin Eye Hospital, Tianjin, China, approved this school-based cohort study (No: 2022018).
Sampling Method: Probability Sample
Enrollment: 34400 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
changes of sphere | change from baseline at 36 months
  changes of sphere
changes of cylinder | change from baseline at 36 months
  changes of cylinder
changes of spherical equivalent | change from baseline at 36 months
  changes of spherical equivalent
changes and distribution of visual acuity | change from baseline at 36 months
  changes and distribution of visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, director, Study Chair — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

REFERENCES:
- [Background] Hu Y, Zhao F, Ding X, Zhang S, Li Z, Guo Y, Feng Z, Tang X, Li Q, Guo L, Lu C, Yang X, He M. Rates of Myopia Development in Young Chinese Schoolchildren During the Outbreak of COVID-19. JAMA Ophthalmol. 2021 Oct 1;139(10):1115-1121. doi: 10.1001/jamaophthalmol.2021.3563. PMID 34529002
- [Background] Ma D, Wei S, Li SM, Yang X, Cao K, Hu J, Fan S, Zhang L, Wang N. Progression of myopia in a natural cohort of Chinese children during COVID-19 pandemic. Graefes Arch Clin Exp Ophthalmol. 2021 Sep;259(9):2813-2820. doi: 10.1007/s00417-021-05305-x. Epub 2021 Jul 21. PMID 34287693